CLINICAL TRIAL: NCT04325958
Title: The Influence of Age on Driving-related Cannabis Effects: Exploring Cannabis Use Frequency and Related Factors
Brief Title: Age Differences in the Effects of Cannabis on Simulated Driving
Acronym: ADCUF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 048/2019
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Cannabis
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: Participants will complete a session with active cannabis and a session with placebo cannabis.
  Order of sessions is randomized.
  Participants and Investigator are blinded.
  Allocation to arms is not randomized. Arms are based on their age.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Age group 19 to 25 (Other): Participants will complete two sessions: one where they drive the simulator before and after smoking a placebo cannabis cigarette (<1% THC), the other where they drive the simulator before and after smoking an active cannabis cigarette (15% ± 5% THC).
  Interventions: Drug: Cannabis; Drug: Placebos
- Age group 35 to 45 (Other): Participants will complete two sessions: one where they drive the simulator before and after smoking a placebo cannabis cigarette (<1% THC), the other where they drive the simulator before and after smoking an active cannabis cigarette (15% ± 5% THC).
  Interventions: Drug: Cannabis; Drug: Placebos

INTERVENTIONS:
Drug: Cannabis — 750mg cigarette of plant material
  Other Names: Marijuana
Drug: Placebos — 750mg cigarette of plant material
  Other Names: Dummy

SUMMARY:
Epidemiological studies suggest that the use of cannabis is associated with an increase in the risk of motor vehicle collisions. It is also known that younger users may be at increased risk for motor vehicle collisions. Further, the frequency with which cannabis is used may be an important variable in determining the effects of cannabis on driving. The purpose of the present study will be to investigate the effects of cannabis on simulated driving in young as compared to middle-aged drivers. Half of the participants will be occasional users of cannabis and half will be frequent users of cannabis.

DETAILED DESCRIPTION:
Epidemiological studies have established that the use of cannabis can increase the risk of a motor vehicle collision. A number of variables can influence the effects of cannabis on driving. For example, frequent users of cannabis have been shown to have different cognitive and physiological responses to cannabis as compared to occasional users. In addition, we know that younger drivers are more likely to be involved in motor vehicle collisions after alcohol use as compared to older users. The contribution of age and experience with cannabis on cannabis-mediated effects on driving have yet to be delineated in laboratory studies. The purpose of the present investigation will be to determine whether cannabis has different effects on driving in young, as compared to middle aged, drivers. Half of each age group will be occasional users of cannabis and the other half will be frequent users.

Eligible participants will attend the laboratory for two test sessions; in one session they will smoke a cannabis cigarette and in the other they smoke a placebo cigarette. Participants will drive a driving simulator before and after smoking the cigarette. Blood for measurement of THC and metabolites will also be collected before smoking the cigarette and at a number of times after smoking. Subjective and cognitive tasks will be completed before and after smoking.

It is hoped that the findings of this study will help to inform public perception and policy into the potential effects of cannabis on driving.

ELIGIBILITY:
Inclusion Criteria

* 19-25 or 35-45 years of age;
* Use of smoked cannabis at least once in the past 6 months.
* Use of smoked or vaped cannabis primarily for recreational purposes on up to 1 day per week or on at least 6 days per week in the past 3 months;
* Holds a class G or G2 Ontario driver's licence (or equivalent from another jurisdiction) for at least 12 months;
* Willing to abstain from using alcohol for 24 hours and cannabis for 72 hours prior to Practice and Test Sessions;
* Willing to abstain from all other drugs not prescribed for medical purposes for 48 hours prior to Practice and Test Sessions;
* Resides within Toronto (study site) or can reside with friends/family in Toronto after a Test Session; this area may be extended to the Greater Toronto area if recruitment challenges arise;
* Participant willing to use appropriate contraception until their participation in the study is completed;
* Provides written and informed consent.

Exclusion Criteria

* Use of cannabis primarily for therapeutic purposes, or equally for therapeutic and recreational purposes;
* Diagnosis of medical condition that contraindicates use of cannabis determined by self-report as judged by the Principal Investigator and a study physician; this includes a history of hypersensitivity to cannabinoids smoke, respiratory disease and/or severe cardiovascular, cerebrovascular, renal or liver disease, and bleeding disorders. Smoking cannabis is not recommended for individuals with respiratory diseases, and they will be excluded;
* Diagnosis of psychiatric condition that contraindicates use of cannabis determined by self-report or SCID-5;
* Participants of childbearing potential: Pregnancy (point-of-care test) or breastfeeding;
* Meets criteria for current or lifetime alcohol or other substance use disorder (DSM-5), except tobacco use disorder and caffeine use disorder;
* Is a regular user of medications that affect brain function (based on self-report); this includes concomitant therapy with sedative-hypnotics or other psychoactive drugs
* Use of anti-hypertensives;
* First-degree relative diagnosed with schizophrenia or another psychotic disorder.
* Participation in a past driving study at CAMH (to limit practice effects).
* Participation in a clinical study concurrent with their participation in this study.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Standard deviation of lateral position | Before cannabis exposure and 30 minutes and 2 hours after cannabis exposure
  A measure of 'weaving' when driving the simulator (meters)

SECONDARY OUTCOMES:
Mean speed | Before cannabis exposure and 25 minutes and 2 hours after cannabis exposure
  A measure of the average speed while driving the simulator (km/hr)
Standard deviation of speed | Before cannabis exposure and 25 minutes and 2 hours after cannabis exposure
  A measure of the variability in speed while driving the simulator (km/hr)
Maximum speed | Before cannabis exposure and 25 minutes and 2 hours after cannabis exposure
  A measure of the greatest speed obtained while driving the simulator (in km/hr)
Following distance | Before cannabis exposure and 25 minutes and 2 hours after cannabis exposure
  A measure of the distance between the car being driven and the car in front (meters)
Braking latency | Before cannabis exposure and 25 minutes and 2 hours after cannabis exposure
  A measure of the time it takes to move the foot from the gas pedal to the brake when a stop sign is encountered (seconds)
Number of collisions | Before cannabis exposure and 25 minutes and 2 hours after cannabis exposure
  The number of collisions while driving the simulator (total number)
Blood concentration of delta-9-tetrahydrocannabinol (THC) | Before cannabis exposure and 25 minutes and 2 hours after cannabis
  A measure of the psychoactive component of cannabis in blood (ng/ml)
Blood concentration of carboxy-tetrahydrocannabinol (THC-COOH) | Before cannabis exposure and 25 minutes and 2 hours after cannabis
  A measure of the inactive metabolite of cannabis in blood (ng/ml)
Blood concentration of 11-hydroxy-tetrahydrocannabinol (11-OH-THC) | Before cannabis exposure and 25 minutes and 2 hours after cannabis
  A measure of the active metabolite of cannabis in blood (ng/ml)
Systolic blood pressure | Before cannabis exposure and 5, 15, 25 minutes and 1, 2, 3, 4 and 5 hours after cannabis
  A vital sign (mmHg)
Diastolic blood pressure | Before cannabis exposure and 5, 15, 25 minutes and 1, 2, 3, 4 and 5 hours after cannabis
  A vital sign (mmHg)
Heart rate | Before cannabis exposure and 5, 15, 25 minutes and 1, 2, 3, 4 and 5 hours after cannabis
  A vital sign (beats/minute)
Visual Analog Scales such as 'I feel this effect', 'I like this drug effect', 'I feel the good effects' | Before cannabis exposure and 5, 15, 25 minutes and 1, 2, 3, 4 and 5 hours after cannabis
  A measure of the subjective effects of cannabis (on a scale of 0 to 100, where is 100 is the strongest level of agreement)
Trail Making Test | Before cannabis exposure and 70 minutes after cannabis
  A measure of the cognitive effects of cannabis (performance speed in seconds)
Verbal Free Recall Task | Before cannabis exposure and 70 minutes after cannabis
  A measure of the cognitive effects of cannabis (number correct)
Grooved Pegboard Test | Before cannabis exposure and 70 minutes after cannabis
  A measure of the cognitive effects of cannabis (performance speed in milliseconds)
Simple and Choice Reaction Time Tasks | Before cannabis exposure and 70 minutes after cannabis
  A measure of the cognitive effects of cannabis (milliseconds)
Vienna Risk-Taking Test | One hour after cannabis exposure
  A measure of the amount of risk-taking (latency)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Wickens, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No